CLINICAL TRIAL: NCT04222907
Title: The Relationship Between GBS Screening in Pregnant Women Insured in Maccabi Healthcare Services (MHS) and Early-onset Neonatal Disease in Israel
Status: Completed | Type: Observational
Sponsor: Assuta Hospital Systems (Other)
Responsible Party: Sponsor
Other Study IDs: 0008-17
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2017-04

CONDITIONS: Streptococcal Infection Group B as Cause of Diseases Classified Elsewhere (Diagnosis)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 20 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women screened for GBS: All women who were pregnant during 2015-2016 and delivery was between 37-42 weeks who were screened for GBS during pregnancy
- Women not screened for GBS: All women who were pregnant during 2015-2016 and delivery was between 37-42 weeks who were not screened for GBS during pregnancy

SUMMARY:
Determination of GBS colonization rates in Pregnant Women insured with Maccabi Health Services, Doctors' Compliance Rates for Referral for Testing, test execution rates, and Early-onset GBS Disease (EOGBSD) Rates in Israel. Determine the relationship between conducting a GBS test in pregnant women and EOGBSD in Israel.

DETAILED DESCRIPTION:
There have been few studies in recent years, which has prompted us to undertake this study. Our aim was to examine the current colonization rates and attack rates in the Israeli population. Our secondary aim was to evaluate the need to readjust recommendations towards universal screening.

ELIGIBILITY:
Inclusion Criteria:

* All women with term pregnancies from 2015 to 2016 (until 20/9/16) insured by Maccabi Healthcare Services (MHS)

Exclusion Criteria:

* repeat pregnancies occurring in the same woman during the time period
* multiple pregnancies
* gestational age greater than 42 weeks due to probability of data inaccuracy
* women with missing information

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Full-term pregnancies were defined as gestational age 37 weeks and above. Pregnancies were identified by a pregnancy code accessed by the primary physician indicating that the patient is pregnant, open pregnancy record in the medical record or child linked to the mother's id. Gestational age was defined by last menstrual period (LMP) or first obstetric ultrasound if LMP was unknown.We identified and excluded repeat pregnancies occurring in the same woman during the time period, multiple pregnancies, gestational age greater than 42 weeks due to probability of data inaccuracy and women with missing information.
Sampling Method: Non-Probability Sample
Enrollment: 54759 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-09-20 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Attack rate of early-onset GBS disease (EOGBSD) | 2015-2016
  Attack rate of (EOGBSD)